CLINICAL TRIAL: NCT03339349
Title: Weight-Based Enoxaparin Dosing and Real-Time Dose Adjustment in Orthopaedic Trauma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 102526
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolus
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enoxaparin Metabolism (Experimental): Eligible patients will have steady state peak and trough anti-Xa levels drawn after the third enoxaparin dose. For patients in-range (levels 0.2-0.4 IU/mL), no intervention will be undertaken. For patients out of range, enoxaparin dose will be adjusted according to an established dose adjustment algorithm. Repeat levels will be checked after the third administration of the new dose.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Enrolled patients will receive real-time monitoring of peak and trough steady state anti-Xa levels. Out-of-range patients will receive real time dose adjustment of Enoxaparin using a clinical protocol developed with our inpatient pharmacists.

SUMMARY:
The rates of Venous thromboembolism (VTE) after orthopedic surgery are as high as 40-60% without prophylactic measures. Enoxaparin, a low-molecular-weight heparin, produces an anticoagulant effect by binding antithrombin, thereby accelerating antithrombin's inactivation of coagulation factor Xa (FXa), thus decreasing the likelihood of clot formation. Despite standard dosing enoxaparin prophylaxis, VTE rates in post-operative orthopedic trauma patients remain as high as 12.2%.The investigators will examine enoxaparin pharmacokinetics and test whether a clinical protocol for real-time enoxaparin dose adjustment can favorably alter the proportion of patients with in-range anti-Factor Xa (aFXa) levels. Outcomes will include peak and trough steady-state aFXa levels in response to standard and escalated doses of enoxaparin and the incidence of venous thromboembolism and bleeding events post-surgery. In the trauma and orthopaedic populations, patients with low initial aFXa levels are significantly more likely to develop deep venous thrombosis. Thus, this study has important implications for appropriate enoxaparin dose magnitude and frequency, and may ultimately help to decrease the substantial morbidity and mortality associated with post-operative VTE.

ELIGIBILITY:
Inclusion Criteria:

* Receiving orthopedic trauma surgery
* Able to have enoxaparin initiated within 36 hours after procedure

Exclusion Criteria:

* Intracranial bleeding/stroke
* bleeding disorder
* heparin-induced thrombocytopenia
* creatinine clearance < 30 mL/minute
* epidural catheter
* serum creatinine > 1.6 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enoxaparin Metabolism
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enoxaparin Metabolism
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 80
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolism Events
Description: Any symptomatic venous thromboembolism events, including deep venous thrombosis or pulmonary embolus occurring within 90 days of surgery
Time Frame: 90 days
Population: Only 17 participants reached full 90-day follow up
  Protocol section, "Statistical Methods, Data Analysis and Interpretation," Using an alpha of 0.05 and beta of 0.9, we would need 107 patients to effectively power a similar change for peak aFXa levels in the proposed study. To allow for attrition, we would require n = 137.
Measure: Count of Participants; unit: Participants
Arm/Group | Enoxaparin Metabolism
Number analyzed (Participants) | 17
Participants | 1

2. Primary Outcome: Number of Participants With Bleeding Events
Description: Bleeding events requiring alteration in the course of care within 90 days of surgery
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Enoxaparin Metabolism
Number analyzed (Participants) | 17
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from post-operative day one or two while admitted to the hospital and 90 days post-operative.
Description: Patients will be contacted via telephone or certified letter at 90 days after surgery to identify Venous thromboembolism (VTE) or bleeding complications that were diagnosed or managed at other institutions.
Arm/Group | Enoxaparin Metabolism
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 1/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoxaparin Metabolism (N=80)
Splenic Embolization (Surgical and medical procedures) | 1 (1) — splenic embolization post op day 7 while on enoxaparin

LIMITATIONS AND CAVEATS:
Our recruitment resulted in inadequate power to analyze the data. Using an alpha of 0.05 and beta of 0.9, 107 subjects were needed for effective power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03339349/Prot_SAP_000.pdf